CLINICAL TRIAL: NCT00393965
Title: Phase 1 Open Label, Dose Escalating, Multiple Dose Study to Determine the Safety, Tolerability, Maximum Tolerated Dose, and Pharmacokinetics of MPC-6827 Administered IV Weekly X 3, Repeated Every 28 Days, in Subjects With Refractory Brain Metastases
Brief Title: Multiple Dose Study of MPC-6827 in Subjects With Refractory Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Margaret Yu, MD / Director of Clinical Research, Myriad Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPC-6827-04-002
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-02

CONDITIONS: Brain Neoplasms
Keywords: Metastases; Refractory; Brain
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — verubulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MPC-6827 — 2-hour IV infusion given once weekly for 3 consecutive weeks on a 28-day cycle.

SUMMARY:
Phase 1, Multiple dose Study of MPC-6827 in Subjects with Refractory Brain Metastases.

ELIGIBILITY:
Inclusion Criteria:

* Refractory Brain Metastases
* At least 1 measurable intracranial lesion as defined by RECIST
* ECOG less than or equal to 1
* Adequate hematology/organ function
* No baseline peripheral or central neuropathy above grade 1

Exclusion Criteria:

* Hypersensitivity to Cremophor EL
* Pregnant or Lactating
* Spinal Cord Compression
* Pre-existing dementia/cognitive disfunction
* Require Neupogen or Neulasta to Maintain Neutrophil Count
* Have Primary Brain Cancer
* Have History of Ischemic Heart Disease
* Have Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-12; Primary Completion 2007-08 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 year
Pharmacokinetics | 1 year

SECONDARY OUTCOMES:
Antitumor Activity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Yu, MD, Study Director — Myrexis Inc.
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States